CLINICAL TRIAL: NCT06133478
Title: Double-blind, Placebo-controlled, Ascending Single- and Multiple- Dose Study of the Safety, Tolerability, and Pharmacokinetics of NUV001 Administered Orally to Healthy Adult Participants
Brief Title: Study of the Safety, Tolerability, and Pharmacokinetics of NUV001 Administered Orally to Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nuvamid SA (Industry)
Collaborators: Medpace, Inc. (Industry); LGD (Industry); Anapharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NUV 001-CLI-001
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers
Keywords: Phase 1; Single ascending dose (SAD); Multiple ascending dose (MAD); Safety; Tolerance; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NUV001 active (Experimental): Single oral administration (treatment period 1 - SAD) and after a washout of at least 5 days, repeated once daily (q.d.) administrations for 14 days (treatment period 2 - MAD)
  Interventions: Drug: NUV001 active cohort 1; Drug: NUV001 active cohort 2; Drug: NUV001 active cohort 3; Drug: NUV001 active cohort 4
- NUV001 Placebo (Placebo Comparator): Single oral administration (treatment period 1 - SAD) and after a washout of at least 5 days, repeated once daily (q.d.) administrations for 14 days (treatment period 2 - MAD)
  Interventions: Drug: NUV001 placebo cohort 1; Drug: NUV001 placebo cohort 2; Drug: NUV001 placebo cohort 3; Drug: NUV001 placebo cohort 4

INTERVENTIONS:
Drug: NUV001 active cohort 1 — 6 participants will be assigned to receive active treatment
  Other Names: NUV001 A mg
  Arms: NUV001 active
Drug: NUV001 active cohort 2 — 6 participants will be assigned to receive active treatment
  Other Names: NUV001 B mg
  Arms: NUV001 active
Drug: NUV001 active cohort 3 — 6 participants will be assigned to receive active treatment
  Other Names: NUV001 C mg
  Arms: NUV001 active
Drug: NUV001 active cohort 4 — 6 participants will be assigned to receive active treatment
  Other Names: NUV001 D mg
  Arms: NUV001 active
Drug: NUV001 placebo cohort 1 — 2 participants will be assigned to receive placebo
  Arms: NUV001 Placebo
Drug: NUV001 placebo cohort 2 — 2 participants will be assigned to receive placebo
  Arms: NUV001 Placebo
Drug: NUV001 placebo cohort 3 — 2 participants will be assigned to receive placebo
  Arms: NUV001 Placebo
Drug: NUV001 placebo cohort 4 — 2 participants will be assigned to receive placebo
  Arms: NUV001 Placebo

SUMMARY:
This blinded placebo-controlled study is designed to evaluate the safety, tolerability, and PK in healthy participants of a single- and multiple-doses (SAD and MAD) of a new investigational drug: NUV001

DETAILED DESCRIPTION:
This is a phase I, single-center, double blind, randomized, single- and multiple-dose, study in four (4) cohorts of eight (8) healthy adult male and female participants per period and dose level.

This study is designed to evaluate the safety, tolerability, and PK in healthy participants of a single- and multiple-doses (SAD and MAD) of a new investigational drug: NUV001

The study will consist of a screening period up to 28 days followed by two (2) treatment periods per participant:

* Treatment Period 1: Single ascending dose (SAD) part with a 3-days inpatient period.
* Treatment Period 2: Multiple ascending dose (MAD) part with a 16-days inpatient period. Dosing from Period 2 Day 1 to Day 14.

A washout of at least 5 days after the first dosing (Period 1 Day 1) should take place between the two periods. A follow-up visit will take place between 6 to 10 days after last dosing (i.e., D14 in period 2) or early discontinuation.

NUV001 will be given orally at four dose levels. Each participant will undergo two treatment periods, but they will receive only one dose level.

The decision to proceed to subsequent dosing cohorts will be made based on a blinded review of the emerging safety data and available PK data.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy all the following inclusion criteria before being allowed to enter the study:

1. Male or female 18 to 55 years of age inclusive, at screening.
2. A body mass index (BMI) between 18.00 and 30.00 kg/m² inclusive and a body weight between 60 kg and 100 kg for males (inclusive), and 50 kg and 100 kg for females (inclusive).
3. Healthy as determined by the investigator based on medical history, physical examination findings, clinical laboratory test results, and digital 12 lead ECG readings (all results should be normal or, if out of range, non-clinically significant as determined by the Investigator).
4. Vital signs at Screening and Admission are within the following ranges:

   * Systolic blood pressure 90-140 mmHg (inclusive);
   * Diastolic blood pressure 50-90 mmHg (inclusive);
   * Heart rate 40-100 beats per minute (inclusive);
   * Oral temperature 36.0-37.5°C (inclusive);
5. AST, ALT, and Total bilirubin are <1.5 x ULN Screening and Admission.
6. Serum creatinine is <1.5 mg/dL and estimated glomerular filtration rate is ≥60 mL/min/1.73 m2 based on Chronic Kidney Disease Epidemiology Collaboration at Screening and Admission.
7. QTcF is ≤450 ms for males and ≤470 ms for females at Screening and Admission.
8. Non-smoker and no use of tobacco or nicotine-containing products for 6 months prior to screening.
9. Have a high probability for compliance with and completion of the study.
10. Female participants of childbearing potential [meaning who are not either surgically sterile (bilateral tubal ligation/occlusion, bilateral salpingectomy, bilateral oophorectomy or hysterectomy) or post-menopausal (no spontaneous menstrual periods for at least two years), confirmed by serum follicle stimulating hormone [FSH] in post-menopausal range based on laboratory reference range, must commit to using a highly effective method of birth control and throughout the entire study and for 90 days after last dose of study drug:

    1. Combined hormonal estrogen and progestogen-containing, or progestogen-only hormonal contraception associated with inhibition of ovulation, started at least 4 weeks prior to the dosing and condom with spermicide for the male partner.
    2. Intrauterine device or intrauterine hormone-releasing system placed at least 4 weeks prior to the dosing, and condom with spermicide for the male partner.
    3. Simultaneous use of a diaphragm or cervical cap with intravaginally applied spermicide and, for the male partner, a male condom with spermicide.
    4. Sterile male partner, i.e., vasectomized since at least 3 months before dosing.
    5. Female participants with same-sex or no partner (when in line with the preferred and usual subject's lifestyle) must agree to use an acceptable form of birth control for duration noted above if they were to become sexually active with a male partner. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.

    NB: Surgically sterile women, if the surgery (bilateral tubal ligation/occlusion, bilateral salpingectomy, bilateral oophorectomy, or hysterectomy) was performed at least 3 months prior to dosing, and female participants who have same-sex sexual relations do not have to use contraception. If the surgery was performed less than 3 months before dosing, the female subject will be considered a woman of childbearing potential (WOCBP).
11. Male participants with a female partner of childbearing potential will be required to be vasectomized at least 3 months prior to screening or use a condom with spermicide throughout the duration of the study and for 90 days after last dose of study drug.
12. Male participants with same-sex or no partner (when in line with the subject's preferred and usual lifestyle) must agree to use an acceptable form of birth control for duration noted above if they were to become sexually active with a female partner of childbearing potential.
13. Agree to avoid sperm or egg donation during the study and for 90 days following last dose of study drug.
14. Can provide a voluntary written informed consent to participate in the study prior to any initiation of study-related procedures.
15. Participant is not subject to any of the following procedures: ward of court, trusteeship, supervision order.

Exclusion Criteria:

If any of the following exclusion criteria apply, the participant must not enter in the study:

Medical History

1. Any significant cardiovascular (e.g., heart failure), hepatic, renal, respiratory (e.g., asthma), gastrointestinal, endocrine (e.g., diabetes, dyslipidemia), immunologic, dermatological, hematological, neurologic, psychiatric disease or history of any clinically important drug allergy.
2. Acute disease state (e.g., vomiting, fever, diarrhea) within 7 days before Day 1 of Treatment Period 1 (SAD).
3. Pregnant or lactating female.
4. Inability to follow study procedures.
5. Use of recreational drugs within 1 year before Day 1 of Treatment Period 1 (SAD).
6. History of alcoholism within 1 year before Day 1 of Treatment Period 1 and/or Regular alcohol consumption >14 units of alcohol per week (1 unit = ½ pint [approximately 240 mL] beer, 25 mL of 40% spirit or a 125 mL glass of wine) within 3 months prior to the admission.
7. Donation of blood or blood loss (i.e., > 400 mL) within 90 days before Day 1 of Treatment Period 1 (SAD).
8. Known allergy or intolerance to study drug, or excipients present in drug product.

   Physical and Laboratory Findings
9. Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibody at Screening.
10. Positive findings of urine drug screen [methadone, barbiturates, oxycodone, amphetamines, methamphetamines, opiates, cannabinoids, cocaine, benzodiazepines, tricyclic antidepressants (TCA), 3,4-methylenedioxy-methamphetamine (MDMA; ecstasy), phencyclidine, cotinine] at screening or admission.
11. Positive Covid -19 by rapid antigen test at admission.

    Prohibited Treatments and study restrictions:
12. Use of any investigational drug within 30 days before study drug administration on Day 1 of Treatment Period 1 (SAD) except for medications needed to treat Adverse Events.
13. Use of prescription or over the counter (OTC) medications, herbal supplements, antacids, vitamins, minerals or food supplements (especially those containing tryptophane, vitamin B3 (NAM and niacin)) within the previous 14 days or 5 half-lives (whichever is longer) before Day 1 of Treatment Period 1 (SAD) and throughout the study and follow-up visit (except for occasional use of nonsteroidal anti-inflammatory drugs (NSAIDs) or acetaminophen, and oral contraception for females of childbearing potential).
14. Consumption of grapefruit juice, alcoholic beverages or any caffeine-containing products or stimulating beverages containing xanthine derivatives (e.g., coffee, tea, chocolate, or soda) for 48 hours prior to dosing on D1 until D2 (Treatment Period 1 (SAD)) and for 48 hours prior to dosing on D1 until the end of the inpatient period (for Treatment Period (MAD)).
15. Participants will be requested to abstain from strenuous physical activity, for 4 days prior to D1 of each treatment period (SAD/MAD), during confinement for each treatment period and 4 days prior to the follow up visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Safety as measured by subject incidence of treatment-emergent adverse events (SAD/MAD) | SAD: First dose date (treatment period 1 Day 1) plus 1 day (until discharge), MAD: First dose date (treatment period 2 Day 1) up to discharge (treatment period 2 Day 15) plus 10 days (follow up visit).
  Percentage of Participants Who Experienced Any Adverse Events.
Safety as measured by subject incidence of treatment-emergent clinically significant changes in vital signs (SAD/MAD) | SAD: First admission (treatment period 1 Day -1) until discharge (treatment period 1 Day 2); MAD: Second admission (treatment period 2 Day -1) up to discharge (treatment period 2 Day 15) plus 10 days (follow up visit).
  Subject incidence of treatment-emergent clinically significant changes in vital signs (Systolic and Diastolic Blood Pressure in millimeters of mercury (mmHg), Heart Rate in beats per minute (bpm), and Oral Body temperature in Celsius).
Safety as measured by subject incidence of treatment-emergent clinically significant changes in Electrocardiograms (SAD/MAD) | SAD: First admission (treatment period 1 Day -1) until discharge (treatment period 1 Day 2); MAD: Second admission (treatment period 2 Day -1) up to discharge (treatment period 2 Day 15) plus 10 days (follow up visit).
  Subject incidence of treatment-emergent clinically significant changes in 12-lead ECGs (PR interval in milliseconds (msec), QRS duration in milliseconds (msec), QRS axis in milliseconds (msec), QT interval in milliseconds (msec)).
Safety as measured by subject incidence of treatment-emergent clinically significant changes in Blood safety tests (SAD/MAD) | SAD: First admission (treatment period 1 Day -1) until discharge (treatment period 1 Day 2); MAD: Second admission (treatment period 2 Day -1) up to discharge (treatment period 2 Day 15) plus 10 days (follow up visit).
  Subject incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests (Complete Blood Count (absolute counts and %), Fasting blood glucose concentration and Serum concentrations in Electrolytes, Protein, Albumin, Total Bilirubin, Blood urea nitrogen, Creatinine, Aspartate Aminotransferase, Alanine Aminotransferase, estimated Glomerular Filtration Rate (eGFR using CKD EPI equation, Activated partial thromboplastin time (aPTT) and Prothrombin Time test (PT) with International Normalized Ratio (INR)).
Safety as measured by subject incidence of treatment-emergent clinically significant changes in Urinalysis safety tests (SAD/MAD) | SAD: First admission (treatment period 1 Day -1) until discharge (treatment period 1 Day 2); MAD: Second admission (treatment period 2 Day -1) up to discharge (treatment period 2 Day 15) plus 10 days (follow up visit).
  Subject incidence of treatment-emergent clinically significant changes in Urinalysis safety tests (pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, and leukocyte esterase).
Safety as measured by subject incidence of treatment-emergent clinically significant changes in Weight (SAD/MAD) | SAD: First admission (treatment period 1 Day -1) until discharge (treatment period 1 Day 2); MAD: Second admission (treatment period 2 Day -1) up to discharge (treatment period 2 Day 15) plus 10 days (follow up visit).
  Subject incidence of treatment-emergent clinically significant changes in Weight in kilograms (Kg).

SECONDARY OUTCOMES:
NUV001 concentration in whole blood (SAD/MAD) | Treatment period 1 (SAD) : Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after dosing on Day 1; Treatment period 2 (MAD) : Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after dosing on Days 1 and 14 and Predose on Days 4, 8 and 12
  Evolution from baseline of NUV001 concentration in whole blood
NUV001 metabolite A concentration in whole blood (SAD/MAD) | Treatment period 1 (SAD) : Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after dosing on Day 1; Treatment period 2 (MAD) : Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after dosing on Days 1 and 14 and Predose on Days 4, 8 and 12
  Evolution from baseline of NUV001 metabolite A concentration in whole blood
NUV001 metabolite B concentration in plasma (SAD/MAD) | Treatment period 1 (SAD) : Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after dosing on Day 1; Treatment period 2 (MAD) : Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after dosing on Days 1 and 14 and Predose on Days 4, 8 and 12
  Evolution from baseline of NUV001 metabolite B concentration in plasma
NUV001 metabolite C concentration in plasma (SAD/MAD) | Treatment period 1 (SAD) : Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after dosing on Day 1; Treatment period 2 (MAD) : Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours after dosing on Days 1 and 14 and Predose on Days 4, 8 and 12
  Evolution from baseline of NUV001 metabolite C concentration in plasma
NUV001 metabolite C concentration in urine (SAD/MAD) | Treatment period 1 (SAD) : collection at Predose and during intervals 0-6, 6-12 and 12-24 hours on Day 1 ; Treatment period 2 (MAD) : collection at Predose and during intervals 0-6, 6-12 and 12-24 hours on Days 1 and 14
  Evolution from baseline of NUV001 metabolite C concentration in urine
NUV001 metabolite D concentration in urine (SAD/MAD) | Treatment period 1 (SAD) : collection at Predose and during intervals 0-6, 6-12 and 12-24 hours on Day 1 ; Treatment period 2 (MAD) : collection at Predose and during intervals 0-6, 6-12 and 12-24 hours on Days 1 and 14
  Evolution from baseline of NUV001 metabolite D concentration in urine

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Brune, MD, Principal Investigator — Medpace, Inc.
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No